- 1 STATISTICAL ANALYSIS PLAN ENDOSCRATCH
- 2 TRIAL NCT03108157

3

- 4 Study title:
- 5 Endometrial Scratch Effect on Pregnancy Rates in Patients Undergoing Egg-donation
- 6 IVF

7

- 8 ClinicalTrials.gov ID:
- 9 NCT03108157
- 10 Version
- 11 25th July 2019
- 12 Protocol Version
- 2.0 2nd November 2016 (1.PROTOCOLO SCRATCH V 2.0.docx.pdf)
- 14 Data Collection Form Version
- 15 1.0 2nd November 2016 (2. CRD.pdf)

16 Signatures

| Principal investigator | SAP author | SAP reviewer |
|------------------------|------------|---------------------|
| Alexandra Izquierdo | David Lora | Alexandra Izquierdo |

17 Note: Add name, surname and date next to the signature.

# 18 SAP reviews

19

| Protocol<br>Version | SAP review | Section<br>modified | Description<br>and reason for<br>modification | Date of modification |
|---|---|---|---|---|

# 1 Introduction

- 22 1.1 Background
- 23 Embryo implantation remains one of the main challenges in assisted reproduction.
- 24 Relevant improvements have been accomplished in reproductive medicine: different
- 25 protocols for controlled ovarian stimulation and endometrial preparation, embryo culture
- with time-lapse technologies, embryo pre-implantational genetic testing and endometrial
- 27 genetic assessment for implantation potential. Despite the fact that these changes have
- 28 led to increasing pregnancy rates in the last few years, the implantation process is still
- 29 inefficient, as it remains around 30% of all embryos replaced (1), and it is not yet totally
- 30 understood.

3132

21

## 1.2 Study justification

- 33 Several studies have tried to determine whether an endometrial injury performed in the
- 34 cycle preceding the embryo transfer in in vitro fertilization (IVF) cycles could enhance
- embryo implantation. Barash et al (2) reported for the first time a two-fold increase in
- 36 pregnancy rate in patients that had undergone multiple ES before the IVF cycle, compared
- 37 to those patients who had no ES performed.
- 38 Since then, many authors have tried to determine ES effects after controlled ovarian
- 39 stimulation (COS), but while some of them have found an increase in pregnancy rates (2–
- 40 5), many others have been unable to find such differences (6–11). The main limitation in
- reaching a conclusion is that most of these are underpowered observational studies, with
- 42 a low number of patients included, with differences in timing (luteal or follicular phase
- from the preceding or same cycle), number of ES (one, two or more procedures), type of
- catheter and different stimulation protocols. It is important to note that those studies that
- 45 have found some positive effects of ES have included patients with implantation failures
- 46 (5,12) whereas those that included patients in their first or second IVF cycle were unable
- 47 to find any differences (8,9). It is also relevant that some studies included as control
- patients, those who had undergone a hysteroscopy prior to the IVF cycle and, even if an
- 49 ES was not performed in these patients, we may assume that the endometrium was
- exposed to some "damage" as well (13). Another study included a cervical biopsy for
- 51 those patients included in the control group, what cannot be really considered as
- 52 "placebo" (10).

- A systematic review conducted by Potdar et al (14) including 7 studies with 2062 patients,
- found a three-fold increase in pregnancy rates in those patients that received ES. Similar
- results were also found some time later by a Cochrane Review by Nastri et al (15) with
- 56 moderate-quality evidence, signaling the need for well-designed trials without uterine
- 57 instrumentation in the control group, stratification for implantation failure and the
- 58 necessity to report live birth rates. This review also showed that endometrial injury on the
- day of oocyte retrieval decreased live birth (RR 0.31, 95% CI 0.14 to 0.69) and clinical
- 60 pregnancy (RR 0.36, 95% CI 0.18 to 0.71).
- All these studies were conducted after COS, but there is only one retrospective study in
- 62 patients receiving embryos from donor eggs, and who have not undergone ovarian
- stimulation (14). When comparing egg donation cycles to other IVF treatments, we find
- two main differences: the first one is that embryo quality is presumably optimal, since all
- embryos come from donor eggs, avoiding the confusion factor of embryo quality
- according to maternal issues (age, BMI, polycystic ovaries, low ovarian reserve...) and
- 67 the second difference is that all patients receive hormone replacement therapy with a
- 68 homogeneous preparation of the endometrium, avoiding different hormonal
- 69 environments caused by diverse responses to controlled ovarian stimulation in IVF.

### 70 1.3 Implantation Failure

- 71 Embry implantation is a complex process that requires successive coordinated steps to
- allow the embryo attach and invade the inner layers of the endometrium.
- 73 Implantation failure definition is very heterogeneous. Coughlan et al (17) considered
- 74 implantation failure if 4 or more good quality embryos had been replaced in 2 or more
- 75 embryo transfers.
- When there is a suspicion of implantation failure, it is necessary to perform certain tests
- in order to exclude possible causes: embryo genetic testing, maternal coagulation and
- 78 immune problems and window of implantation determination and thus endometrial
- 79 receptivity to the embryo.
- 80 The endometrium is a dynamic tissue with a complex architecture that undergoes several
- 81 changes during the menstrual cycle which have an important impact on embryo
- 82 implantation. Endometrial scratching (ES) is a simple procedure aiming to create a mild

- 83 endometrial injury that has been proposed to improve the embryo-endometrium dialogue.
- 84 Different authors have attributed this improvement to the effects of different cytokines
- and growth factors involved in an acute endometrial inflammatory process (18), the
- 86 enhancement of new vascularization and decidualization (19), the improvement of
- 87 endometrial maturation (13), and the promotion of endometrial gene expression that may
- lead to a better synchrony between the embryo and the endometrium (20).
- 89 2 Hypothesis, objective and aim of the clinical trial
- 90 2.1 Study hypothesis [level 2]
- Patients that receive ES during the cycle preceding the embryo transfer, have increased
- 92 endometrial receptivity and thus higher clinical pregnancy rates (CPR).
- 93 2.1.1 Operative hypothesis [level 3]
- Null hypothesis: Clinical pregnancy rate in patients who have undergone an ES in the
- previous cycle is not different from those who have not received it.
- Alternative hypothesis: Patients who receive an ES in the previous cycle have a 15%
- 97 higher CPR than those who have not received it.
- 98 2.2 Main outcome [level 2]
- 99 The main objective of the ENDOSCRATCH trial is to determine if there are differences
- in pregnancy rates in egg donor IVF treatments when comparing patients receiving an ES
- before endometrial preparation for embryo transfer and those who will not receive any
- intervention. CPR will be determined by the visualization of a intrauterine gestational sac
- via vaginal ultrasound at approximately 6 weeks pregnancy.
- 104 2.2.1 Secondary outcomes [level 3]
- 105 2.2.1.1 Efficacy secondary outcomes [level 4]
- 1. Secondary endpoints are biochemical pregnancy rate (BPR), ongoing pregnancy
- rate (OPR), implantation rate (IR), miscarriage rate (MR), live birth rate (LBR)
- and cumulative pregnancy rate (CumPR).
- a. Biochemical pregnancy rate will be determined by the ratio between the
- number of patients with blood β-hCG levels over 10 mUI/ml 12 days after

| 111 | the emotyo transfer and the number of emotyo transfers. |
|---|---|
| 112 | b. Ongoing pregnancy will be assessed via ultrasound beyond 12 weeks of |
| 113 | pregnancy. |
| 114 | c. Implantation rate will be determined by the ratio between the number of |
| 115 | gestational sacs and the number of replaced embryos. |
| 116 | d. Miscarriage rate will be determined by the ratio between the number of |
| 117 | miscarriages and the total number of pregnancies. |
| 118 | Early miscarriage will be assessed if pregnancy stops before the 12 <sup>th</sup> week |
| 119 | of pregnancy. Late miscarriage will be assessed if pregnancy stops |
| 120 | between the 12 <sup>th</sup> and the 24 <sup>th</sup> week of pregnancy. |
| 121 | e. Live birth rate will be determined by the ratio between babies born and the |
| 122 | number of embryo transfers. |
| 123 | f. Multiple pregnancy rate, determined by the ratio between the number of |
| 124 | multiple pregnancies and the total number of pregnancies. |
| 125 | g. CumPR will be evaluated 12 months after randomization for all patients. |
| 126 | 2. To determine the possible beneficial effect of ES in egg donor IVF recipients |
| 127 | adjusted by: age, BMI, smoking habits. |
| 128 | 3. To evaluate the CPR in both groups regarding the donor's age, male partner's age |
| 129 | and sperm quality, number of eggs obtained and fertilized, total number of |
| 130 | embryos obtained and quality and number of transferred embryos. |
| 131 | 4. To determine the possible positive effect in specific treatment subgroups: |
| 132 | a. Previous implantation failures from IVF with own eggs |
| 133 | b. Previous implantation failures from IVF with donor eggs |
| 134 | c. Previous miscarriages |
| 135 | d. Previous live births |
| 136 | 5. To evaluate the interference of ES with the endometrial preparation, in terms of: |
| 137 | a. Endometrial thickness |
| 138 | b. Stimulation duration |
| 139 | c. Dose of medication needed |
| 140 | |

the embryo transfer and the number of embryo transfers.

111

| 141 | 2.2.1.2 Safety secondary outcomes [level 4] |
|---|---|
| 142<br>143 | 1. Obstetric outcome analysis to evaluate the possible association of this technique with: |
| 144 | a. Early or late miscarriage |
| 145 | b. Placentation anomalies |
| 146 | c. Intrauterine growth restriction |
| 147 | d. Preterm birth |
| 148 | e. Premature membrane rupture |
| 149 | f. Gestational diabetes |
| 150 | g. Gestational hypertension |
| 151 | 2. Secondary effects of ES: |
| 152 | a. Pain |
| 153 | b. Bleeding |
| 154 | 3 Clinical trial design [level 1] |
| 155 | 3.1 Clinical trial description [level 2] |
| 156 | This is a single-centre prospective RCT, fully conducted at ProcreaTec Fertility Clinic in |
| 157 | Madrid, starting January 2017 to December 2019 to evaluate the effectiveness of an |
| 158 | endometrial biopsy (scratching) before endometrial preparation, during the luteal phase |
| 159 | of the previous cycle versus the conventional treatment protocol for egg donation IVF |
| 160 | without endometrial biopsy. |
| 161 | 3.1.1 Clinical trial summarized description [level 3] |
| 162 | 1. Study: Interventional. |
| 163 | 2. Assignment: Randomized. |
| 164 | 3. Final classification: Efficacy study. |
| 165 | 4. Intervention model: Parallel assignment. |
| 166 | 5. Blinding: Not blinded. |
| 167 | 6. Main outcome: The improvement in clinical pregnancy rate in egg donor IVF |
| 168 | recipients. |

## 169 3.2 Patient randomization [level 2]

- 170 Patients starting egg donor IVF cycles that fulfill inclusion criteria will be offered
- participation. If they agree they will be assigned to a treatment group according to the
- 172 randomization chart, which will be obtained by a web-based randomization program
- using random blocks (randomization.com). Since patients in the study group will receive
- an intervention and those in the control group will not (no placebo intervention will be
- performed), blinding is not possible for patients nor for physicians. All patients will sign
- 176 IC to be enrolled in the study.
- 1. Group A (176 patients): Intervention group. They will receive an ES during the
- luteal phase of the previous cycle to embryo transfer.
- 2. Group B (176 patients): Control group. They will undergo the conventional
- protocol for donor IVF treatment.
- 181 3.3 Sample size calculation [level 2]
- The average CPR after embryo transfer in egg donor IVF cycles is 60% at our centre.
- Based on previous studies, where the difference in CPR for IVF cycles varied between
- 184 10 to 30%(2,4,5,12,14,21-23), we estimated that a 15% difference in CPR would be
- clinically relevant. According to that percentage, a total of 332 patients will be needed to
- detect a 15% difference between the two groups, with 80% statistical power and two-
- sided alpha of 0,05. Considering a 5% dropout rate, we will include 176 patients per study
- arm, 352 patients in total.
- 189 3.4 Interim analysis [level 2]
- 190 Non applicable.
- 191 3.5 Study setting [level 2]
- We will collect data from patients undergoing an egg donor IVF cycle at ProcreaTec
- 193 Fertility Centre in Madrid from the 13th of January 2017.
- 194 3.5.1 Eligible population [level 2]
- 195 Those patients undergoing an egg donor IVF treatment protocol will be eligible for this
- 196 study.

- 197 3.5.2 Study population [level 2]
- 198 Study population will include those patients fulfilling the inclusion criteria who have
- accepted the study and signed the IC.
- 200 3.5.3 Inclusion and exclusion criteria
- 201 3.5.3.1 Inclusion criteria:
- 202 Patients will be included if they meet the following inclusion criteria:
- 203 Age between 18 and 50 years
- 204 Primary or secondary infertility
- 205 Patients undergoing an IVF protocol with donor eggs
- 206 Normal uterine cavity (transvaginal ultrasound scan)
- 207 Patients with endometrial polyps can be included as long as polypectomy is performed
- at least two months before the treatment cycle
- 209 3.5.3.2 Exclusion criteria:
- 210 Patients will be excluded if:
- 211 There is a severe male factor (less than 2 million sperms per ml)
- 212 They have uterine anomalies such as uterine fibroids that impact the cavity, Mullerian
- 213 malformations or severe adenomyosis
- 214 They have unilateral or bilateral hydrosalpinx
- 215 They have undergone a previous ES or hysteroscopy (at least one month before the
- 216 randomization)
- 217 Pre-implantation genetic testing cycles
- 218 3.6 Data collection
- All study variables will be collected from patients included in the trial, from ProcreaTec
- 220 clinical records, according to the information required in the data collection form (Annex
- 221 I). Each doctor will include relevant information in the patients' clinical record and the
- 222 principal investigator will be responsible for collecting and managing the information.
- 223 Any adverse events will be reported by responsible doctors and managed by the principal
- investigator.

- 225 3.7 Ethical approval [level 2]
- 226 This study will be conducted after the authorization of the Ethical Committee of Princesa
- 227 Hospital in Madrid (Registry nº 2934/12-01-2017). Clinical data will be treated
- confidentially following the Spanish data protection law (Spanish Organic Law 15/1999,
- 229 13<sup>th</sup>Dec).
- 230 4 Statistical principles [level 1]
- 231 4.1 General considerations
- 232 Baseline characteristics of patients included will be analyzed as follows. Qualitative
- variables will be described using mean and standard deviation, non-normal variables will
- be summarized using median and 25% and 75% centiles. Qualitative variables will be
- 235 described using frequency distribution.
- The main outcome, CPR, and secondary outcomes, BPR, OPR, MR, IR, LBR and CumPR
- for each group will be analyzed with Chi-Squared test or Fisher's exact test. Efficacy of
- 238 the treatment will be described as absolute and relative frequencies, together with the
- association strength by raw risk ratio (RR) with 95% confidence intervals. In addition, a
- 240 general linear model, with a log link and binomial distribution, will be used to estimate
- 241 the strength of association between primary and secondary outcomes adjusted by
- independent variables.
- Results will be presented as RR and 95% confidence intervals. Statistical significance
- will be 0.05 (5% both sides  $\alpha$  error) for all comparisons. Statistical analysis will be done
- using Stata 13 for Windows (StataCorp LP, Texas).
- All analyses will be performed by the 9th version of SAS system.
- 247 4.2 Study population [level 2]
- 248 The main statistical analysis will be by intention to treat (ITT). Patients allocated to a
- determined treatment group will be followed and evaluated as members of that group,
- without regards to the fulfillment of the planned treatment.
- 251 4.3 Patient flow diagram [level 2]
- 252 Patient diagram flow will be detailed with the CONSORT standards (fig 1).



Figure 1. CONSORT patient flow diagram.

#### 4.4 Outcome evaluation

# 4.4.1 Efficacy outcome

The primary study objective will be to evaluate if endometrial scratching improves CPR in patients undergoing egg-donation IVF versus patients without endometrial scratching. The primary study objective will be performed using the Chi-square statistic test at a 2-sided significance level of alpha = 0.05. The intervention effect will be quantified using the risk ratio (RR) with the 95% confidence interval and p-value (). The RR estimation will be realized using a generalized regression model with log link and binary outcome (clinical pregnancy equal to yes or no). The intervention RR will be adjusted by the following pre-treatment variables (Tabl): age, BMI, smoker, previous live birth, previous biochemical miscarriage, previous miscarriage, number of previous failed cycles with own eggs. Also, a multivariate model with the treatment will be performed to predict the CPR (Table 4). Finally, a predictive model will be generated with the treatment and the previous covariables.

| | Group A<br>(n=XXX) | Group B<br>(n=XXX) | RR (IC 95%) | p-value |
|---|---|---|---|---|
| Biochemical pregnancy | NN (X%) | NN (X%) | XX (XX;XX) | P=XX |
| Clinical pregnancy | NN (X%) | NN (X%) | XX (XX;XX) | P=XX |
| Ongoing pregnancy | NN (X%) | NN (X%) | XX (XX;XX) | P=XX |
| Early miscarriage | NN (X%) | NN (X%) | XX (XX;XX) | P=XX |
| Late miscarriage | NN (X%) | NN (X%) | XX (XX;XX) | P=XX |
| Abortion | NN (X%) | NN (X%) | XX (XX;XX) | P=XX |
| Live birth | NN (X%) | NN (X%) | XX (XX;XX) | P=XX |
| Multiple pregnancy | NN (X%) | NN (X%) | XX (XX;XX) | P=XX |
| Cumulative clinical pregnancy rate (12 months) | NN (X%) | NN (X%) | XX (XX;XX) | P=XX |

278 Table 1. Clinical outcome

| | GROUP A (n=XXX) | GROUP B<br>(n=XXX) |
|---|---|---|
| Race | | |
| Arabian | XX (X%) | XX (X%) |
| Asian | XX (X%) | XX (X%) |
| Caucasian | XX (X%) | XX (X%) |
| Mixed | XX (X%) | XX (X%) |
| Hispanic | XX (X%) | XX (X%) |
| Mulatto | XX (X%) | XX (X%) |
| Black | XX (X%) | XX (X%) |
| Age | XX(XX) | XX (XX) |
| BMI | XX (XX) | XX (XX) |
| Smoking habit | XX (X%) | XX (X%) |
| Previous live birth | XX (X%) | XX (X%) |
| Previous miscarriage | XX (X%) | XX (X%) |
| Previous biochemical miscarriage | XX (X%) | XX (X%) |
| Previous ectopic pregnancy | XX (X%) | XX (X%) |
| Previous abortion | XX (X%) | XX (X%) |
| Number of previous failed cycles with own eggs | | |
| 0 | XX (X%) | XX (X%) |
| 1 | XX (X%) | XX (X%) |
| 2 | XX (X%) | XX (X%) |
| +2 | XX (X%) | XX (X%) |
| Number of previous failed cycles with donor eggs | | |
| 0 | XX (X%) | XX (X%) |
| 1 | XX (X%) | XX (X%) |
| 2 | XX (X%) | XX (X%) |
| +2 | XX (X%) | XX (X%) |

Table 2. Baseline characteristics

| | Group A<br>(n=XXX) | Group B<br>(n=XXX) | p-value |
|---|---|---|---|
| Donor's age | NN (X%) | NN (X%) | P=XX |
| Male partner's age | NN (X%) | NN (X%) | P=XX |
| Fresh sperm | NN (X%) | NN (X%) | P=XX |
| Frozen sperm | NN (X%) | NN (X%) | P=XX |
| Donor sperm | NN (X%) | NN (X%) | P=XX |
| Total sperm count | NN (X%) | NN (X%) | P=XX |
| Number of MII obtained | NN (X%) | NN (X%) | P=XX |
| Number of fertilized eggs | NN (X%) | NN (X%) | P=XX |
| Total number of embryos obtained | NN (X%) | NN (X%) | P=XX |
| Number of replaced embryos | NN (X%) | NN (X%) | P=XX |
| Quality of replaced embryos | | | |
| HATCHED | NN (X%) | NN (X%) | P=XX |
| HATCHING | NN (X%) | NN (X%) | P=XX |
| EXPANDED | NN (X%) | NN (X%) | P=XX |
| EARLY BLASTOCYST | NN (X%) | NN (X%) | P=XX |
| MORULA | NN (X%) | NN (X%) | P=XX |
| CLEAVAGE STAGE | NN (X%) | NN (X%) | P=XX |

280 Table 3. Cycle characteristics

| Adjusted model | | |
|----------------------------------|-------------|---------|
| | RR (CI 95%) | p-value |
| Group A vs Group B | XX (XX;XX) | P=XX |
| Age | XX (XX;XX) | P=XX |
| Group A vs Group B | XX(XX;XX) | P=XX |
| BMI | XX(XX;XX) | P=XX |
| Group A vs Group B | XX (XX;XX) | P=XX |
| Smoking habit | XX (XX;XX) | P=XX |
| Group A vs Group B | XX (XX;XX) | P=XX |
| Previous live births | XX (XX;XX) | P=XX |
| Group A vs Group B | XX (XX;XX) | P=XX |
| Previous biochemical miscarriage | XX (XX;XX) | P=XX |
| Group A vs Group B | XX (XX;XX) | P=XX |
| Previous miscarriage | XX (XX;XX) | P=XX |
| Group A vs Group B | XX (XX;XX) | P=XX |
| Previous IVF own-eggs | XX (XX;XX) | P=XX |
| Group A vs Group B | XX (XX;XX) | P=XX |
| Previous IVF donor eggs | XX (XX;XX) | P=XX |

Table 4. Model to evaluate the CPR and LBR according with the treatment and adjusted by age, BMI, smoking habit, previous live birth, previous biochemical miscarriage, previous miscarriage, previous IVF own eggs or previous IVF donor eggs failures.

| Multivariate model | | |
|---|---|---|
| RR (CI 95%) p-value | | |
| <b>Endometrial scratching vs no intervention</b> | XX (XX;XX) | P=XX |
| Age | XX (XX;XX) | P=XX |
| BMI | XX (XX;XX) | P=XX |
| Smoking habit | XX (XX;XX) | P=XX |
| Previous live birth | XX (XX;XX) | P=XX |
| Previous biochemical pregnancies | XX (XX;XX) | P=XX |
| Previous miscarriages | XX (XX;XX) | P=XX |
| Previous failed own eggs IVF embryo transfers | XX (XX;XX) | P=XX |
| Previous failed egg-donor IVF embryo transfers | XX (XX;XX) | P=XX |

Table 5. Multivariate model to evaluate the CPR with the treatment adjusted by covariables

285

286

The following subgroups for the CPR will be defined (Table 6): previous implantation failures with own eggs, previous implantation failures with donor eggs, previous

miscarriage, previous live births. In each group, the effect of endometrial scratching (RR) for the CPR will be estimated using a generalized lineal model with log link and binary outcome (CPR equal yes or no). The comparison between groups will be realized using interaction between treatment and subgroup in the generalized linear model.

| | GROUP A | | GROUF | B | |
|---|---|---|---|---|---|
| | CPR | Total | CPR | Total | RR (IC 95%) |
| Previous implantation failures with own eggs (p=XX) | | | | | |
| Yes | XX (XX%) | XX | XX (XX%) | XX | XX (XX;XX) |
| No | XX (XX%) | XX | XX (XX%) | XX | XX (XX;XX) |
| Previous implantation failures with donor eggs (p=XX) | | | | | |
| Yes | XX (XX%) | XX | XX (XX%) | XX | XX (XX;XX) |
| No | XX (XX%) | XX | XX (XX%) | XX | XX (XX;XX) |
| Previous<br>miscarriages<br>(p=XX) | | | | | |
| Yes | XX (XX%) | XX | XX (XX%) | XX | XX (XX;XX) |
| No | XX (XX%) | XX | XX (XX%) | XX | XX (XX;XX) |
| Previous live births (p=XX) | | | | | |
| Yes | XX (XX%) | XX | XX (XX%) | XX | XX (XX;XX) |
| No | XX (XX%) | XX | XX (XX%) | XX | XX (XX;XX) |

Table 6. Effect of endometrial scratching on CPR by subgroups

The effect of endometrial scratching on secondary study objectives, LBR and CumPR, will be evaluate using the Chi-square statistic test at a 2-sided significance level of alpha = 0.05. The intervention effect will be quantified using the risk ratio (RR) with the 95% confidence interval and p-value (). The RR estimation will be realized using a generalized regression model with log link and binary outcome (clinical pregnancy equal to yes or no). The intervention RR will be adjusted by the following pre-treatment variables (Tabl): age, BMI, smoker, previous live

birth, previous biochemical miscarriage, previous miscarriage, number of previous failed cycles with own eggs and donor eggs.

The effect of endometrial scratching on stimulation duration, endometrial thickness and total dose required will be evaluate using the Student's t statistic test at a 2-sided significance level of alpha = 0.05. If the normality hypothesis is not rejected with the Shapiro-Wilk test, the objective variables will be presented using the mean and the standard deviation. If the normality hypothesis is rejected, the variables will be analyzed with no-parametric test of Mann-Whitney and summarized with the median and range interquartile, 25 and 75 percentile. The data will be described according to the Table 7.

| | GROUP A<br>(n=XXX) | GROUP B<br>(n=XXX) | p-value |
|---|---|---|---|
| Stimulation duration | XX (XX) | XX (XX) | P=XX |
| <b>Endometrial thickness</b> | XX (XX) | XX(XX) | P=XX |
| <b>Total dose required</b> | XX (XX) | XX (XX) | P=XX |

Table 7. Results of endometrial preparation

### 4.4.2 Safety outcomes

The effect of endometrial scratching on pregnancy complications: miscarriage, placentation anomalies, intrauterine growth restriction, preterm birth, premature membrane rupture, gestational diabetes and gestational hypertension, will be evaluated using the Chi-square statistic test at a 2-sided significance level of alpha = 0.05. The intervention effect will be quantified for each safety outcome using the risk ratio (RR) with the 95% confidence interval and p-value (). The RR estimation will be realized using a generalized regression model with log link and binary outcome (yes or no). The intervention RR will be summarized according to Table 8.

| | GROUP A<br>(n=XXX) | GROUP B<br>(n=XXX) | RR (IC 95%) | p-value |
|---|---|---|---|---|
| Miscarriage | XX (X%) | XX (X%) | XX (XX;XX) | P=XX |
| Placentation abnomalies | XX (X%) | XX (X%) | XX (XX;XX) | P=XX |
| Intrauterine growth restriction | XX (X%) | XX (X%) | XX (XX;XX) | P=XX |
| Preterm birth | XX (X%) | XX (X%) | XX (XX;XX) | P=XX |
| Premature membrane rupture | XX (X%) | XX (X%) | XX (XX;XX) | P=XX |
| Gestational diabetes | XX (X%) | XX (X%) | XX (XX;XX) | P=XX |
| Gestational hypertension | | | | |

319 Table 8. Obstetrical outcome.

323

334

- The absolute and relative frequencies of the pain and bleeding will be summarized by the
- patient with endometrial scratching. The endometrial preparation time will be described
- with the median, range interquartile, 25 and 75 percentile.

#### 4.5 Baseline characteristics

- 324 The baseline characteristics: demographics, clinical, laboratory and relationship with the
- 325 treatments will be presented with the mean and standard deviation values or absolute and
- relative frequency according to the treatment. If the distribution of continuous variable is
- not normal (Kolmogorov-Smirnov test), the information will be summarized with median
- and range interquartile, 25 and 75 percentile.

#### 329 4.6 Evaluation of lost or unknown data.

- The outlier data will be described with the maximum and minimum values. The outlier
- values will be revised with the CRD and corrected it. As loss to follow-up is expected to
- be minimal (i.e. less than one percent missing data on primary and secondary outcomes),
- missing values will not be imputed.

#### 4.7 Additional considerations

- When the fifty percent of the cells have expected counts less than five, the chi-square
- tests will be replaced by Fisher's exact test.

- 337 The protocol or statistical analysis plan deviation will be described and justified in the
- deviation documents.

| 339 | 5 GLOSSARY |
|---|---|
| 340 | BMI: body mass index |
| 341 | BPR: Biochemical pregnancy rate |
| 342 | CI: confidence interval |
| 343 | COS: Controlled ovarian stimulation |
| 344 | CPR: Clinical pregnancy rate |
| 345 | CumPR: Cumulative pregnancy rate |
| 346 | ES: Endometrial scratching |
| 347 | IC: Informed consent |
| 348 | CI: Confidence Interval |
| 349 | IR: implantation rate |
| 350 | IUI: Intrauterine insemination |
| 351 | IVF: In vitro Fertilization |
| 352 | LBR: Live birth rate |
| 353 | MR: miscarriage rate |
| 354 | OPR: ongoing pregnancy rate |
| 355 | OR: Odds ratio |
| 356 | RR: Risk ratio |
| 357 | |
| 358 | 6 REFERENCES |
| 359<br>360 | 1. De Geyter C, Calhaz-Jorge C, Kupka MS, Wyns C, Mocanu E, Motrenko T, et al. ART in Europe, 2014: results generated from European registries by ESHRE: The |

- European IVF-monitoring Consortium (EIM) for the European Society of Human
- Reproduction and Embryology (ESHRE). Hum Reprod Oxf Engl. 2018
- 363 01;33(9):1586–601.
- 364 2. Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the
- 365 endometrium doubles the incidence of successful pregnancies in patients
- undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317–22.
- 367 3. Raziel A, Schachter M, Strassburger D, Bern O, Ron-El R, Friedler S. Favorable
- influence of local injury to the endometrium in intracytoplasmic sperm injection
- patients with high-order implantation failure. Fertil Steril. 2007 Jan;87(1):198–201.
- 370 4. Zhou L, Li R, Wang R, Huang H, Zhong K. Local injury to the endometrium in
- 371 controlled ovarian hyperstimulation cycles improves implantation rates. Fertil Steril.
- 372 2008 May;89(5):1166–76.
- 373 5. Karimzadeh MA, Ayazi Rozbahani M, Tabibnejad N. Endometrial local injury
- improves the pregnancy rate among recurrent implantation failure patients
- undergoing in vitro fertilisation/intra cytoplasmic sperm injection: a randomised
- 376 clinical trial. Aust N Z J Obstet Gynaecol. 2009 Dec;49(6):677–80.
- 6. Frantz S, Parinaud J, Kret M, Rocher-Escriva G, Papaxanthos-Roche A, Creux H,
- et al. Decrease in pregnancy rate after endometrial scratch in women undergoing a
- first or second in vitro fertilization. A multicenter randomized controlled trial. Hum
- 380 Reprod Oxf Engl. 2019 Jan 1;34(1):92–9.
- 381 7. Lensen S, Osavlyuk D, Armstrong S, Stadelmann C, Hennes A, Napier E, et al. A
- Randomized Trial of Endometrial Scratching before In Vitro Fertilization. N Engl J
- 383 Med. 2019 24;380(4):325–34.
- 384 8. Yeung TWY, Chai J, Li RHW, Lee VCY, Ho PC, Ng EHY. The effect of
- endometrial injury on ongoing pregnancy rate in unselected subfertile women
- undergoing in vitro fertilization: a randomized controlled trial. Hum Reprod Oxf
- 387 Engl. 2014 Nov;29(11):2474–81.
- 388 9. Eskew AM, Reschke LD, Woolfolk C, Schulte MB, Boots CE, Broughton DE, et al.
- 389 Effect of endometrial mechanical stimulation in an unselected population
- undergoing in vitro fertilization: futility analysis of a double-blind randomized
- controlled trial. J Assist Reprod Genet. 2018 Nov 5;
- 392 10. Baum M, Yerushalmi GM, Maman E, Kedem A, Machtinger R, Hourvitz A, et al.
- Does local injury to the endometrium before IVF cycle really affect treatment
- outcome? Results of a randomized placebo controlled trial. Gynecol Endocrinol Off
- 395 J Int Soc Gynecol Endocrinol. 2012 Dec;28(12):933–6.
- 396 11. Gibreel A, El-Adawi N, Elgindy E, Al-Inany H, Allakany N, Tournaye H.
- Endometrial scratching for women with previous IVF failure undergoing IVF
- 398 treatment. Gynecol Endocrinol Off J Int Soc Gynecol Endocrinol. 2015
- 399 Apr;31(4):313–6.
- 400 12. Nastri C, Ferriani R, Raine-Fenning N, Martins W. Endometrial scratching 401 performed in the non-transfer cycle and outcome of assisted reproduction: a

- randomized controlled trial. Ultrasound Obstet Gynecol. 2013;42(4):375-382.
- 403 13. Nastri CO, Lensen S, Polanski L, Raine-Fenning N, Farquhar CM, Martins WP.
- Endometrial injury and reproductive outcomes: there's more to this story than meets
- the horse's blind eye. Hum Reprod Oxf Engl. 2015 Mar;30(3):749.
- 406 14. Potdar N, Gelbaya T, Nardo LG. Endometrial injury to overcome recurrent embryo
- implantation failure: a systematic review and meta-analysis. Reprod Biomed Online.
- 408 2012 Dec;25(6):561–71.
- 409 15. Nastri CO, Lensen SF, Gibreel A, Raine-Fenning N, Ferriani RA, Bhattacharya S,
- et al. Endometrial injury in women undergoing assisted reproductive techniques.
- Cochrane Database Syst Rev [Internet]. 2015 [cited 2019 Jun 7];(3). Available from:
- https://www.cochranelibrary.com/cdsr/doi/10.1002/14651858.CD009517.pub3/full
- ?highlightAbstract=reproduct%7Cwoman%7Cin%7Cwithdrawn%7Cundergoing%
- 414 7Cinjuri%7Creproductive%7Ctechniqu%7Cassisted%7Cendometrial%7Ctechniqu
- es%7Cendometri%7Creproductiv%7Cassist%7Cinjury%7Cundergo%7Cwomen
- 416 16. Dain L, Ojha K, Bider D, Levron J, Zinchenko V, Walster S, et al. Effect of local
- 417 endometrial injury on pregnancy outcomes in ovum donation cycles. Fertil Steril.
- 418 2014 Oct;102(4):1048–54.
- 419 17. Coughlan C, Ledger W, Wang Q, Liu F, Demirol A, Gurgan T, et al. Recurrent
- 420 implantation failure: definition and management. Reprod Biomed Online. 2014
- 421 Jan;28(1):14–38.
- 422 18. Cakmak H, Taylor HS. Implantation failure: molecular mechanisms and clinical
- 423 treatment. Hum Reprod Update. 2011 Apr;17(2):242–53.
- 424 19. Gnainsky Y, Granot I, Aldo PB, Barash A, Or Y, Schechtman E, et al. Local injury
- of the endometrium induces an inflammatory response that promotes successful
- 426 implantation. Fertil Steril. 2010 Nov;94(6):2030–6.
- 427 20. Kalma Y, Granot I, Gnainsky Y, Or Y, Czernobilsky B, Dekel N, et al. Endometrial
- biopsy-induced gene modulation: first evidence for the expression of bladder-
- transmembranal uroplakin Ib in human endometrium. Fertil Steril. 2009
- 430 Apr;91(4):1042–9, 1049.e1-9.
- 431 21. Narvekar SA, Gupta N, Shetty N, Kottur A, Srinivas M, Rao KA. Does local
- endometrial injury in the nontransfer cycle improve the IVF-ET outcome in the
- subsequent cycle in patients with previous unsuccessful IVF? A randomized
- controlled pilot study. J Hum Reprod Sci. 2010 Jan;3(1):15–9.
- 435 22. Seval MM, Şükür YE, Özmen B, Kan Ö, Sönmezer M, Berker B, et al. Does adding
- endometrial scratching to diagnostic hysteroscopy improve pregnancy rates in
- women with recurrent in-vitro fertilization failure? Gynecol Endocrinol Off J Int
- 438 Soc Gynecol Endocrinol. 2016 Dec;32(12):957–60.
- 439 23. Maged AM, Rashwan H, AbdelAziz S, Ramadan W, Mostafa WAI, Metwally AA,
- et al. Randomized controlled trial of the effect of endometrial injury on implantation
- and clinical pregnancy rates during the first ICSI cycle. Int J Gynaecol Obstet Off
- 442 Organ Int Fed Gynaecol Obstet. 2018 Feb;140(2):211–6.